CLINICAL TRIAL: NCT05084573
Title: Continuous Standard Bupivacaine Interscalene Block Versus Single Injection Liposomal Bupivacaine Following Surgical Fixation of Proximal Humerus Fractures
Brief Title: Continuous Interscalene Block vs Liposomal Bupivacaine After Proximal Humerus Fracture Surgery
Acronym: CLIP-H
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Chi-Wing, Honorary Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 20-247
Record Dates: First submitted 2021-01-21; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Shoulder Fractures
Keywords: interscalene nerve block; shoulder surgery
MeSH Terms: conditions — Shoulder Fractures | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to receive either continuous interscalene nerve block (CISB) using standard bupivacaine OR a single interscalene injection of liposomal bupivacaine (LB).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects, investigators, and all parties involved in patient management or data collection will be blinded throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine (Experimental): Patients will receive a single bolus interscalene injection of 10mL 1.33% LB followed by placement of indwelling (sham) catheter in the interscalene region. Upon arrival in the recovery room, a nurse will connect the catheter to a fixed-rate portable elastometric pump (Easypump®, B Braun, Germany) filled with 300mL normal saline (NS) at a default fixed rate of infusion of 5mL/hr. The syringe, catheter, pump and clamp will be covered by opaque black bags to conceal the milky appearance of LB. The catheter will be removed on postoperative day 2.
  Interventions: Drug: Liposomal bupivacaine
- Standard bupivacaine CISB (Active Comparator): Patients will receive a single bolus interscalene injection of 10mL 0.25% SB followed by placement of indwelling (sham) catheter in the interscalene region. Upon arrival in the recovery room, a nurse will connect the catheter to a fixed-rate portable elastometric pump (Easypump®, B Braun, Germany) filled with 300mL 0.2% SB at a default fixed rate of infusion of 5mL/hr. The syringe, catheter, pump and clamp will be covered by opaque black bags to conceal the drug appearance. The catheter will be removed on postoperative day 2.
  Interventions: Drug: Standard bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Single bolus injection 10mL 1.33% LB
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Standard bupivacaine — Single bolus 10mL 0.25% SB + continuous 300mL 0.2% SB @5mL/hr
  Other Names: Marcaine; Sensorcaine
  Arms: Standard bupivacaine CISB

SUMMARY:
The purpose of this study is to compare the efficacy of continuous interscalene block (CISB) using standard bupivacaine versus a single interscalene injection of liposomal bupivacaine (LB) on pain control following surgical fixation of proximal humerus fractures.

DETAILED DESCRIPTION:
Restricted range of motion following open reduction and internal fixation (ORIF) of proximal humerus fractures is a potential complication that severely limits functional outcomes . It must therefore be avoided by adequate pain control in order to allow for early mobilisation in addition to physiotherapy.

Interscalene block (ISB) is one of the most effective and widely used regional analgesic options shoulder surgeries. ISB can be delivered as a single injection or by continuous infusion via an indwelling catheter. While continuous interscalene block (CISB) offers a longer duration of analgesia as compared to a single injection of the same anaesthetic, it carries an inherent risk of catheter malposition, dislodgement, and infection.

As compared to standard bupivacaine (SB), liposomal bupivacaine (LB) is a formulation designed to prolong the duration of analgesia up to 72 hours via a single injection. While this could avoid the need for an indwelling catheter, results of studies comparing LB to CISB have been inconsistent.

The purpose of this is non-inferiority trial is to compare the effectiveness of a single injection of LB versus CISB with SB on pain control following ORIF of proximal humerus fractures. The study hypothesis is that LB is not unacceptably worse than CISB with regard to pain control in the first two postoperative days.

Patients providing informed consent will be screened for eligibility. All eligible patients will be randomly assigned in a double-blind manner (participant and investigator) and a 1:1 ratio to receive either LB or CISB.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age between 18 and 80
* Isolated Proximal humeral fracture (AO Types 31.A1-3 and B1-3 or Neer 2/3 part or greater tuberosity fracture equivalent)
* Locking Plate fixation
* Split deltoid minimal invasive approach

Exclusion Criteria:

* Revision surgery
* Impaired cognitive function (Abbreviated Mental Test Score (AMT score) < 8)
* 4 part fractures
* Poor surgical reduction quality
* Unable to attend rehabilitation
* Preexisting shoulder problems
* Fracture fixation stability unable to tolerate early passive motion exercise
* Use of implants other than a locking plate for fracture fixation
* Activity of daily living is dependent on others
* Polytrauma
* Use of deltopectoral approach
* Patient unable to follow post-operative rehabilitation protocol with early mobilization
* Allergy to amide local anaesthetics, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS), opioids
* Respiratory Disease with limited respiratory reserve
* Cardiac Disease: Any degree of Heart Block, Heart Failure
* Neurological: Any Seizure Disorder
* Psychiatric illnesses affecting pain perception e.g. severe depression and anxiety disorder
* Alcohol or substance abuse
* Chronic Pain, other than chronic knee pain
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* Impaired Renal Function (defined as preoperative eGFR < 30ml /min /1.73 m2)
* Impaired Hepatic Function
* Pregnancy
* Inability to use PCA
* Patient refusal to ISB
* Patient refusal to study
* Patients do not understand Cantonese

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain on movement as measured by Numerical Rating Scale (NRS) | At each post-op day 1-7
  Numerical rating scale (NRS) during attempted passive forward shoulder flexion to 90 degrees; 0 points (no pain) to 11 points (worst pain imaginable).
Pain at rest as measured by Numerical Rating Scale (NRS) | At each post-op day 1-7
  Numerical rating scale (NRS) at rest; 0 points (no pain) to 11 points (worst pain imaginable).

SECONDARY OUTCOMES:
Intraoperative opioid consumption | Intraoperative
  Intraoperative IV remifentanil consumption (mcg/kg/min)
Incidence of ISB related complications | Intraoperative to post-op day 3
  Complications related to interscalene block
PCA morphine consumption | From immediately post-operation to post-op day 2
  Amount of patient-controlled analgesia (PCA) morphine consumed (mg)
Number of patients with side effects effects of PCA using morphine | From immediately post-operation to post-op day 2
  Side effects related to opioid use (Nausea/Vomiting, Dizziness, Constipation)
Rescue morphine consumption | From immediately post-operation to post-op day 2
  Additional opioid used in addition to PCA morphine
Total length of stay | Through study completion, an average of 1 year
  Duration of hospital stay (days)
Analgesic consumption after discharge | From post-op day 3 to day 7
  Total analgesic consumption (dihydrocodeine) after hospital discharge (pill count)
Overall Benefit of Analgesia Score (OBAS) | Immediate post-operation to post-op day 3
  Patient-reported measure of pain, side effects, and satisfaction of post-operative analgesia; 7 questions rated from 0 (worst outcome) to 4 (best outcome)
Presence of chronic pain at follow-up | At 2 weeks, 6 weeks and 3 months post-op
  Presence of chronic pain by self-report
Presence of neuropathic pain at follow-up | At post-op 2 weeks, 6 weeks and 3 months
  Presence of neuropathic pain by physical examination and neuropathic pain questionnaire, a 10-item mixed self-report/observer rated physical exam measure ranging from 0 (no pain) to 10, with a score of 4 or greater diagnostic of neuropathic pain
Region-specific physical functioning and symptoms | At post-op 2 weeks, 6 weeks and 3 months
  Physical function and symptoms measured by Shortened Disabilities of the Arm, Shoulder and Hand Questionnaire (QuickDASH), an 11-item patient-reported measure with a total score ranging from 0 (no disability) to 100 (most severe disability).
Health-related quality of life (HRQOL) | At post-op 2 weeks, 6 weeks and 3 months
  12-item Short Form Health Survey (SF-12), a patient-reported outcome measure of HRQOL comprised of a mental component (MCS) and physical component (PCS), each with a final score ranging from 0 (worst outcome) to 100 (best outcome).
Patient satisfaction as measured by the Patient Satisfaction Questionnaire General Satisfaction Subscale | At post-op 2 weeks, 6 weeks and 3 months
  Patient satisfaction with healthcare provision as measured by the Patient Satisfaction Questionnaire General Satisfaction subscale (PSQ18-GS), a two-item subscale with a final score ranging from 0 (lowest satisfaction) to 10 (highest satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wing Chan, Principal Investigator — Queen Mary Hospital, Hong Kong; Christian Xinshuo Fang, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified dataset underlying results to be published as an appendix in final publication.
Supporting Information: Study Protocol, SAP
Time Frame: Aim to publish protocol and analysis plan in a peer-reviewed journal prior to recruitment completion
Access Criteria: Additional information available upon reasonable request of the corresponding author.

REFERENCES:
- [Background] Hodgson SA, Mawson SJ, Stanley D. Rehabilitation after two-part fractures of the neck of the humerus. J Bone Joint Surg Br. 2003 Apr;85(3):419-22. doi: 10.1302/0301-620x.85b3.13458. PMID 12729121
- [Background] Vorobeichik L, Brull R, Bowry R, Laffey JG, Abdallah FW. Should continuous rather than single-injection interscalene block be routinely offered for major shoulder surgery? A meta-analysis of the analgesic and side-effects profiles. Br J Anaesth. 2018 Apr;120(4):679-692. doi: 10.1016/j.bja.2017.11.104. Epub 2018 Feb 13. PMID 29576109
- [Background] Malik O, Kaye AD, Kaye A, Belani K, Urman RD. Emerging roles of liposomal bupivacaine in anesthesia practice. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):151-156. doi: 10.4103/joacp.JOACP_375_15. PMID 28781438
- [Background] Sabesan VJ, Shahriar R, Petersen-Fitts GR, Whaley JD, Bou-Akl T, Sweet M, Milia M. A prospective randomized controlled trial to identify the optimal postoperative pain management in shoulder arthroplasty: liposomal bupivacaine versus continuous interscalene catheter. J Shoulder Elbow Surg. 2017 Oct;26(10):1810-1817. doi: 10.1016/j.jse.2017.06.044. Epub 2017 Aug 24. PMID 28844420
- [Background] Budge M, Orvets N, Shields E. Single-shot liposomal bupivacaine interscalene nerve block provides equivalent pain relief compared to continuous catheter interscalene nerve block in total shoulder arthroplasty. Seminars in Arthroplasty: JSES. 2020;30(4):285-90.
- [Background] Marino J, Scuderi G, Dowling O, Farquhar R, Freycinet B, Overdyk F. Periarticular Knee Injection With Liposomal Bupivacaine and Continuous Femoral Nerve Block for Postoperative Pain Management After Total Knee Arthroplasty: A Randomized Controlled Trial. J Arthroplasty. 2019 Mar;34(3):495-500. doi: 10.1016/j.arth.2018.11.025. Epub 2018 Nov 23. PMID 30583813
- [Background] Weller WJ, Azzam MG, Smith RA, Azar FM, Throckmorton TW. Liposomal Bupivacaine Mixture Has Similar Pain Relief and Significantly Fewer Complications at Less Cost Compared to Indwelling Interscalene Catheter in Total Shoulder Arthroplasty. J Arthroplasty. 2017 Nov;32(11):3557-3562. doi: 10.1016/j.arth.2017.03.017. Epub 2017 Mar 16. PMID 28390888